CLINICAL TRIAL: NCT06598566
Title: A Comparative Evaluation of Nottingham Hip Fracture Score (NHFS) and Acute Physiology and Chronic Health Evaluation (APACHE) II Score to Predict 30-day Mortality in Geriatric Patients Above 60 Years Undergoing Hip Fracture Surgery.
Status: Completed | Type: Observational
Sponsor: Tata Main Hospital (Other)
Responsible Party: Principal Investigator, Dr.Deb Sanjay Nag, HOD & Head Consultant, Anaesthesiology, Tata Main Hospital
Other Study IDs: 2122100200
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Geriatric Hip Fracture
Keywords: Geriatrics; Hip Fractures; APACHE II; Mortality; Morbidity
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Geriatric patients above 60 years undergoing hip fracture surgery: Efficacy of NHFS and APACHE-II in predicting 30-day mortality in geriatric patients above 60 years undergoing hip fracture surgery.
  Interventions: Other: Nottingham Hip Fracture Score (NHFS) score; Other: Acute Physiology and Chronic Health Evaluation (APACHE)-II score

INTERVENTIONS:
Other: Nottingham Hip Fracture Score (NHFS) score — Nottingham Hip Fracture Score (NHFS) score in patients above 60 years undergoing hip fracture surgery.
Other: Acute Physiology and Chronic Health Evaluation (APACHE)-II score — Acute Physiology and Chronic Health Evaluation (APACHE)-II score in patients above 60 years undergoing hip fracture surgery

SUMMARY:
This study aims to compare the Nottingham Hip Fracture Score (NHFS) and the Acute Physiology and Chronic Health Evaluation II (APACHE II) score in predicting 30-day mortality in geriatric patients over 60 years old undergoing hip fracture surgery.

DETAILED DESCRIPTION:
The study aim to compare the Nottingham Hip Fracture Score (NHFS) and the Acute Physiology and Chronic Health Evaluation II (APACHE II) score in predicting 30-day mortality in geriatric patients over 60 years undergoing hip fracture surgery. This study was conducted at the Tata Main Hospital in Jamshedpur, India. The study was designed as a prospective observational study, with data collected from June 2022 to June 2023. The study's primary objective was to predict mortality in patients undergoing hip fracture surgery. The study also investigated secondary outcomes such as the need for postoperative ventilator and ionotropic support, the occurrence of acute kidney injury, cardiac morbidity, and the presence of pulmonary embolism and deep vein thrombosis, as well as length of stay.

ELIGIBILITY:
Inclusion Criteria: Age more than or equal to 60 years, Underwent Hip fracture surgeries, of Either Sex

-

Exclusion Criteria: Age less than 60 years of age, Hip fractures not undergoing any invasive surgery, Implant removals planned for healed hip fractures, Re-explorations during the same admission in which primary surgery was conducted

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted for elective surgery for fractures around the hip joint at at Tata main hospital, Jamshedpur, India
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
  Mortality at least 30 days after surgery or death (during hospital stay or within 30 days after surgery.

SECONDARY OUTCOMES:
Length of Stay (LOS) | 30 days
  Length of Stay (LOS) in the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Tata Main Hospital, Jamshedpur, Jharkhand, India

IPD SHARING:
Plan to Share IPD: Undecided
Being a GDPR compliant organization, data privacy officer's consent may be needed. It has not been taken yet. However, masked data maybe considered if approved by the organization.